CLINICAL TRIAL: NCT05486923
Title: Validity and Reliability Evaluation of the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) for Adult-type Diffuse Gliomas Patients in Chinese Population
Brief Title: Validity and Reliability Evaluation of the PRO-CTCAE for Adult-type Diffuse Gliomas Patients in Chinese Population
Acronym: VERONICA
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jinsong Wu, Chief Physician, Professor, Huashan Hospital
Other Study IDs: KY2022-681
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Glioma; Patient Reported Outcome Measures; Self Report; Adverse Effects
Keywords: Glioma; China; Patient Reported Outcome Measures; Self Report; Humans; Adverse effects; Adult; Surveys and Questionnaires; Research Design
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- KPS less than 70: The patients in this group have Karnofsky performance Status less than 70，and the proportion of them is not less than 15%.
  Patients need regular follow-up surveys within 2 years after the date of surgery.
- KPS more than 70: The patients in this group have Karnofsky performance Status more than 70. Patients need regular follow-up surveys within 2 years after the date of surgery.

SUMMARY:
Given the increasing importance of patient's perspective in adverse events reporting, Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE™) has been proposed as new PRO measures in oncology; however, its implementation has not yet been evaluated in glioma patients, and standardized selection process of priority symptom terms has not been applied.

The study focuses on Chinese adult-type diffuse glioma patients. First, based on information queries, expert consultation research, online Delphi survey, and survey data analysis, the investigators will determine the questionnaire terms for PRO-CTCAE™ for adult-type diffuse gliomas patients. In the next stage, a prospective, multi-center, real-world study to assess the validity, reliability, and responsiveness of the customized PRO-CTCAE™ for adult-type diffuse gliomas patients in Chinese population will be launched (VERONICA).

DETAILED DESCRIPTION:
First, based on information queries, expert consultation research, online Delphi survey, and survey data analysis, the investigators will determine the questionnaire terms for PRO-CTCAE™ for adult-type diffuse gliomas patients.

A total of 16 experts (13 neurosurgeons, 2 radiotherapists, 1 psychiatrist) from 14 medical centers in China were invited to participate in a consensus-seeking 2-round online Delphi survey. Participants rated the level of their agreement with each symptom term likely to occur during adult diffuse gliomas treatment on a 5-point Likert scale. Terms not reaching consensus over the first round were modified in the second rounds. Consensus was defined as content validity index (CVI) >0.78，coefficient of variation (CV)< 0.35 and average Likert score >3.00.

Second, a prospective, multi-center, real-world study would be performed to assess the validity, reliability, and responsiveness of the customized PRO-CTCAE™ for adult diffuse glioma patients in Chinese population.

This study is an observational, prospective, open-label clinical study. It is estimated that 450 adult diffuse glioma patients will be recruited from 17 research centers, and participants will be included in the cohort in chronological order until the target number of cases is reached. The study is expected to be completed within 2 years. In this study, KPS will be used as the anchor point to compare two groups of patients(KPS≤70 and KPS>70, patients with KPS≤70 is not less than 15%).

The investigators do not intervene in the current treatment plan for patients, only observe the treatment plan, and conduct regular questionnaires on the patients: since the patients are enrolled (within 42 days after surgery), six basic follow-ups and long-term follow-ups will be carried out. The whole follow-ups will last for two years.

The follow-up contents include:

Filled out by doctors: demographic information, diagnosis information, anti-tumor treatment (in the past 2 weeks), special treatment (in the past 2 weeks, including but not limited to dehydration drugs and psychotropic drugs, etc.), CTCAE v5.0 (only including the items corresponding to PRO-CTCAE™), KPS.

Filled out by patients: customized PRO-CTCAETM, QLQ-C30, GIC.

Data will be collected using EDC system to ensure patient privacy and data integrity.

The statistical analysis methods:

For the customized PRO-CTCAE™, quantitatively assign each item and its answers (F, S, A, I, P), and then use statistical methods to assess the validity, reliability, and responsiveness of the customized PRO-CTCAE™ for adult diffuse glioma patients in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed adult diffuse glioma patients( including astrocytoma, IDH-mutant; oligodendroglioma, IDH-mutant and1p/19q-codeleted; glioblastoma, IDH-wildtype; other adult diffuse glioma NEC/NOS).
2. For newly diagnosed patients, the patient has not received the first non-surgical treatment.
3. For recurrent patients, the patient has not received the first non-surgical treatment after the recurrence.
4. 18 to 85 years old.
5. No significant cognitive impairment based on researchers' judgment.
6. Patients can use mobile phones or computers on their own or with the help of others, read and understand Chinese, at least with primary school culture.
7. Patients are undergoing anti-tumor treatment and continue to receive treatment within the next 28 days.
8. Patients sign written informed consent.

Exclusion Criteria:

1. Patients who are not considered suitable for this study.
2. Since the diagnosis, the patient has undergone non-surgical treatment.
3. Patients fail to complete the questionnaire within 42 days of signing informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult diffuse glioma patients aged 18 to 85 years who have not received the first non-surgical treatment after diagnosis/recurrent.
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
the validity, reliability, and responsiveness of the customized PRO-CTCAE™ for adult-type diffuse gliomas patients in Chinese population | December 1, 2025
  The investigators will compare the customized PRO-CTCAE™ measurements at multiple visits and test the correlation between PRO-CTCAE™, QLQ-C30 and KPS scores, to access the validity, reliability, and responsiveness of the customized PRO-CTCAE™ for adult-type diffuse gliomas patients in Chinese population.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Wu, Ph.D. & M.D., Study Chair — Huashan Hospital
Locations (14):
- China (14):
  - Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuan Wu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Sanjiu Brain Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Jiangsu People's Hospital, Nanjing, Jiangsu
  - Xijing Hospital, Xi'an, Shaanxi
  - Department of Neurologic Surgery, Huashan Hospital, Shanghai Medical College, Fudan University, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - East Hospital Affiliated To Tongji University, Shanghai, Shanghai Municipality
  - Shanghai Proton and Heavy Ion Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong TS, Dirven L, Arons D, Bates A, Chang SM, Coens C, Espinasse C, Gilbert MR, Jenkinson D, Kluetz P, Mendoza T, Rubinstein L, Sul J, Weller M, Wen PY, van den Bent MJ, Taphoorn MJB. Glioma patient-reported outcome assessment in clinical care and research: a Response Assessment in Neuro-Oncology collaborative report. Lancet Oncol. 2020 Feb;21(2):e97-e103. doi: 10.1016/S1470-2045(19)30796-X. PMID 32007210
- [Background] Basch E, Geoghegan C, Coons SJ, Gnanasakthy A, Slagle AF, Papadopoulos EJ, Kluetz PG. Patient-Reported Outcomes in Cancer Drug Development and US Regulatory Review: Perspectives From Industry, the Food and Drug Administration, and the Patient. JAMA Oncol. 2015 Jun;1(3):375-9. doi: 10.1001/jamaoncol.2015.0530. PMID 26181187
- [Background] Cagney DN, Sul J, Huang RY, Ligon KL, Wen PY, Alexander BM. The FDA NIH Biomarkers, EndpointS, and other Tools (BEST) resource in neuro-oncology. Neuro Oncol. 2018 Aug 2;20(9):1162-1172. doi: 10.1093/neuonc/nox242. PMID 29294069
- [Background] Armstrong TS, Wefel JS, Wang M, Gilbert MR, Won M, Bottomley A, Mendoza TR, Coens C, Werner-Wasik M, Brachman DG, Choucair AK, Mehta M. Net clinical benefit analysis of radiation therapy oncology group 0525: a phase III trial comparing conventional adjuvant temozolomide with dose-intensive temozolomide in patients with newly diagnosed glioblastoma. J Clin Oncol. 2013 Nov 10;31(32):4076-84. doi: 10.1200/JCO.2013.49.6067. Epub 2013 Oct 7. PMID 24101048
- [Background] Gilbert MR, Dignam JJ, Armstrong TS, Wefel JS, Blumenthal DT, Vogelbaum MA, Colman H, Chakravarti A, Pugh S, Won M, Jeraj R, Brown PD, Jaeckle KA, Schiff D, Stieber VW, Brachman DG, Werner-Wasik M, Tremont-Lukats IW, Sulman EP, Aldape KD, Curran WJ Jr, Mehta MP. A randomized trial of bevacizumab for newly diagnosed glioblastoma. N Engl J Med. 2014 Feb 20;370(8):699-708. doi: 10.1056/NEJMoa1308573. PMID 24552317
- [Background] Armstrong TS, Bishof AM, Brown PD, Klein M, Taphoorn MJ, Theodore-Oklota C. Determining priority signs and symptoms for use as clinical outcomes assessments in trials including patients with malignant gliomas: Panel 1 Report. Neuro Oncol. 2016 Mar;18 Suppl 2(Suppl 2):ii1-ii12. doi: 10.1093/neuonc/nov267. PMID 26989127
- [Background] Yeung AR, Pugh SL, Klopp AH, Gil KM, Wenzel L, Westin SN, Gaffney DK, Small W Jr, Thompson S, Doncals DE, Cantuaria GHC, Yaremko BP, Chang A, Kundapur V, Mohan DS, Haas ML, Kim YB, Ferguson CL, Deshmukh S, Bruner DW, Kachnic LA. Improvement in Patient-Reported Outcomes With Intensity-Modulated Radiotherapy (RT) Compared With Standard RT: A Report From the NRG Oncology RTOG 1203 Study. J Clin Oncol. 2020 May 20;38(15):1685-1692. doi: 10.1200/JCO.19.02381. Epub 2020 Feb 19. PMID 32073955
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Basch E, Reeve BB, Mitchell SA, Clauser SB, Minasian LM, Dueck AC, Mendoza TR, Hay J, Atkinson TM, Abernethy AP, Bruner DW, Cleeland CS, Sloan JA, Chilukuri R, Baumgartner P, Denicoff A, St Germain D, O'Mara AM, Chen A, Kelaghan J, Bennett AV, Sit L, Rogak L, Barz A, Paul DB, Schrag D. Development of the National Cancer Institute's patient-reported outcomes version of the common terminology criteria for adverse events (PRO-CTCAE). J Natl Cancer Inst. 2014 Sep 29;106(9):dju244. doi: 10.1093/jnci/dju244. Print 2014 Sep. PMID 25265940
- [Background] Dueck AC, Mendoza TR, Mitchell SA, Reeve BB, Castro KM, Rogak LJ, Atkinson TM, Bennett AV, Denicoff AM, O'Mara AM, Li Y, Clauser SB, Bryant DM, Bearden JD 3rd, Gillis TA, Harness JK, Siegel RD, Paul DB, Cleeland CS, Schrag D, Sloan JA, Abernethy AP, Bruner DW, Minasian LM, Basch E; National Cancer Institute PRO-CTCAE Study Group. Validity and Reliability of the US National Cancer Institute's Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). JAMA Oncol. 2015 Nov;1(8):1051-9. doi: 10.1001/jamaoncol.2015.2639. PMID 26270597
- [Background] Trask PC, Dueck AC, Piault E, Campbell A. Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events: Methods for item selection in industry-sponsored oncology clinical trials. Clin Trials. 2018 Dec;15(6):616-623. doi: 10.1177/1740774518799985. Epub 2018 Sep 19. PMID 30230365